CLINICAL TRIAL: NCT02248168
Title: Mirapex PMS Study Final Report
Brief Title: Post Marketing Surveillance And Special Surveillance for Mirapex® Tablet in Patients With Idiopathic Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.599
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Idiopathic Parkinson's disease patients
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole
  Other Names: Mirapex®

SUMMARY:
The objectives of this study are to investigate issues or questions about MIRAPEX Tablets as shown below through the Post Marketing Surveillance (PMS) study upon approval.

* Unexpected adverse events (especially, serious adverse events (SAEs))
* To find out the status of incidence of adverse events under actual practice
* Factors on the safety profile
* Factors on the efficacy profile

ELIGIBILITY:
Inclusion Criteria:

* Among the patients with idiopathic Parkinson's disease, from those receiving MIRAPEX Tablets first after a contract of the study to the requested number of cases will be consecutively enrolled without skipping

Exclusion Criteria:

* Following patients are contraindicated.

  1. Patients who are hypersensitive to MIRAPEX or its ingredients
  2. Refer to the insert paper for other contraindication.
* Following patients should be carefully administered.

  1. Patient with renal impairment
  2. Refer to the insert paper for other precaution.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with idiopathic Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 1449 (Actual)
Dates: Start 2002-03; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Unified Parkinson's disease Rating Scale (UPDRS) | up to 4 weeks
  Tremor at rest, Rigidity, Body bradykinesia and hypokinesia

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 4 weeks
Global Assessment of efficacy by investigator on 3-point scale | after 4 weeks